CLINICAL TRIAL: NCT02523313
Title: A Phase II Randomized, Double-Blind Trial of Immunotherapy With Nivolumab or Nivolumab Plus Ipilimumab Versus Double-Placebo Control as a Post-Surgical/Post-Radiation Treatment for Stage IV Melanoma With No Evidence of Disease
Brief Title: Immunotherapy With Nivolumab or Nivolumab Plus Ipilimumab vs. Double Placebo for Stage IV Melanoma w. NED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dr. med. Dirk Schadendorf (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Dirk Schadendorf, Prof. Dr. med., University Hospital, Essen
Organization: University Hospital, Essen (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IMMUNED
Record Dates: First submitted 2015-08-05; First posted 2015-08-14 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nivolumab + Placebo (Active Comparator): Nivolumab (3 mg/kg) i.v. every 2 weeks + Placebo instead of Ipilimumab on weeks 1, 4, 7 and 10 + Placebo instead of Nivolumab on weeks 4 and 10
  Interventions: Drug: Nivolumab + Placebo
- Nivolumab + Ipilimumab (Experimental): Nivolumab (1 mg/kg) and Ipilimumab (3 mg/kg) i.v. every 3 weeks for 4 doses. Both study drugs are administered on the same day over the first 12 weeks + Placebo instead of Nivolumab on weeks 3, 5, 9 and 11. After week 12: Nivolumab as maintenance and at a dose of 3 mg/kg IV every 2 weeks for up to 1 year after initial dosing (of the combination) or until PD.
  Interventions: Drug: Nivolumab + Ipilimumab
- Double Placebo Control (Placebo Comparator): Placebo instead of Nivolumab and Placebo instead of Ipilimumab i.v. every 3 weeks for 4 doses. Both placebos are administered on the same day over the first 12 weeks + Placebo instead of Nivolumab on weeks 3, 5, 9 and 11. After week 12 Placebo instead of Nivolumab as maintenance and applied as IV every 2 weeks for up to 1 year after initial dosing (of the combination) or until PD.
  Interventions: Drug: Double Placebo Control

INTERVENTIONS:
Drug: Nivolumab + Placebo — Nivolumab will be applied at a dose of 3 mg/kg given as IV infusion every 2 weeks for up to 1 year after initial dosing or until PD + Placebo instead of Ipilimumab on weeks 1, 4, 7 and 10 + Placebo instead of Nivolumab on weeks 4 and 10.
  Other Names: Treatment Arm A
  Arms: Nivolumab + Placebo
Drug: Nivolumab + Ipilimumab — Nivolumab (1 mg/kg) and Ipilimumab (3 mg/kg) will be applied as IV infusion every 3 weeks for 4 doses. Both study drugs are to be administered on the same day over the first 12 weeks + Nivolumab-Placebo on weeks 3, 5, 9 and 11. After week 12 Nivolumab is given as maintenance and will be applied at a dose of 3 mg/kg IV every 2 weeks for up to 1 year after initial dosing (of the combination) or until PD.
  Other Names: Treatment Arm B
  Arms: Nivolumab + Ipilimumab
Drug: Double Placebo Control — Placebo instead of Nivolumab and Placebo instead of Ipilimumab will be applied as IV infusion every 3 weeks for 4 doses. Both placebos are to be administered on the same day over the first 12 weeks + Placebo instead of Nivolumab on weeks 3, 5, 9 and 11. After week 12 Placebo instead of Nivolumab is given as maintenance and will be applied intravenously every 2 weeks for up to 1 year after initial dosing (of the combination) or until PD.
  Other Names: Treatment Arm C
  Arms: Double Placebo Control

SUMMARY:
This is a prospective, double-blind placebo-controlled, multicenter, randomized phase II trial testing the adjuvant immunotherapy with Nivolumab plus Ipilimumab Placebo or Nivolumab plus Ipilimumab versus Double Placebo Control as a post-surgical/post-radiation treatment for stage IV melanoma with no evidence of disease (NED).

DETAILED DESCRIPTION:
This study will allow for direct comparison of the clinical benefit provided by Nivolumab monotherapy or Nivolumab combined with Ipilimumab versus double placebo control. Furthermore, it will also allow for direct comparison of the respective safety profiles of Nivolumab monotherapy or Nivolumab combined with Ipilimumab. Nivolumab monotherapy was chosen as one of the experimental arms because of a favourable risk-benefit ratio assessed in the large Phase 1 study (MDX1106-03/CA209-003). The combination of Nivolumab and Ipilimumab was chosen as an experimental arm because of the preliminary evidence from the Phase 1 study CA209-004 suggesting synergy between Nivolumab and Ipilimumab resulting in a higher frequency of patients with increased tumour burden reduction. Evaluating both Nivolumab monotherapy and the combination of Nivolumab and Ipilimumab will provide clinical data allowing clinicians to select the appropriate treatment for each patient based on their individual risk-benefit ratio.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV melanoma arising from a primary cutaneous site or metastatic from an unknown primary site with no evidence of disease (NED) after surgery or radiation therapy (conducted within 8 weeks before enrolment)
* Signed written informed consent
* Known BRAF status
* Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
* Minimum life expectancy of five years excluding their melanoma diagnosis
* ECOG performance status of 0 or 1
* Tumor tissue from the resected site of disease must be provided for biomarker analyses. In order to be randomized a subject must have a PD-L 1 expression classification (positive (≥ 5% tumor cells expressing PD-L1) or negative (< 5% tumor cells expressing PD-L1)). If an insufficient amount of tumor tissue from the resected site is provided for analysis, acquisition of additional archived tumor tissue (block and/or slides) for the biomarker analyses is required.
* Prior radiotherapy must have been completed at least 2 weeks prior to study drug administration
* Required laboratory values
* Negative pregnancy test for female subjects and effective contraception (Pearl-Index <1) for both male and female subjects if the risk of conception exists

Exclusion Criteria:

* History of primary uveal or mucosal melanoma
* Prior therapy with CTLA4 or PD1 antibodies
* The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent or to comply with the trial procedures.
* Lack of availability for clinical follow-up assessments.
* Any immunosuppressive therapy given within the past 30 days prior to study drug administration (excluding physiologic steroid hormone replacement)
* Other malignancies within the past five years requiring treatment except basal or squamous skin carcinomas or carcinoma in situ of the cervix
* Serious cardiac, gastrointestinal, hepatic or pulmonary disease reducing life expectancy to less than five years
* Patients with serious intercurrent illness, requiring hospitalization.
* Other serious illnesses, e.g., serious infections requiring antibiotics or bleeding disorders.
* The patient is known to be positive for Human Immunodeficiency Virus (HIV) or other chronic infections (HBV, HCV) or has another confirmed or suspected immunosuppressive or immunodeficient condition.
* Known hypersensitivity reaction to any of the components of study treatment
* Pregnancy (absence to be confirmed by ß-HCG urinary test, minimum sensitivity 25IU/L or equivalent units of HCG)) or lactation period
* Women of childbearing potential (WOCBP): Refusal or inability to use effective means of contraception (Pearl-Index <1). WOCBP will be instructed to adhere to contraception until 31 weeks after the last dose of investigational product
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year (Pearl-Index <1). Men receiving Nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception until 31 weeks after the last dose of investigational product
* Known alcohol or drug abuse
* Participation in another clinical study and use of any investigational or non-registered product (drug or vaccine) within the 30 days before registration
* Significant disease or condition which, in the investigator's opinion, would exclude the patient from the study
* Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2021-06-27 (Actual); Study Completion 2021-06-27 (Actual)

PRIMARY OUTCOMES:
Efficacy of adjuvant immunotherapy with Nivolumab alone or in combination with Ipilimumab (Recurrence-free survival) | 24 months after the last patient ended treatment
  Recurrence-free survival (RFS) defined as the time from date of randomization until the date of the first recurrence (local or distant metastasis), new primary melanoma or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | 24 months after the last patient ended treatment
  The OS of a patient is defined as the time from date of randomization until date of death.
Time to recurrence (TTR) | 24 months after the last patient ended treatment
  The TTR of a patient is defined as the time from date of randomization until date of disease recurrence (local or distant metastasis) or melanoma-related death.
Progression/recurrence free survival 2 (PRFS2) for crossover patients of Arm C | 24 months after the last patient ended treatment
  The PRFS2 is defined as time from date of randomization until the date of first disease progression per RECIST 1.1 beyond the initial unresectable disease recurrence, the date of second recurrence in patients without evidence of disease after surgery of a resectable first recurrence or the date of death, whichever occurs first.

OTHER OUTCOMES:
Safety / Toxicity All adverse events ≥ Grade 3 according to CTCAE Version 4.0 criteria | until 90 days after discontinuation of dosing
  All adverse events ≥ Grade 3 according to CTCAE Version 4.0 criteria, that are related to the administration of the investigational agents will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Schadendorf, Prof. Dr., Principal Investigator — Studienzentrum Hautklinik Universitätsklinikum Essen Klinik f. Dermatologie
Locations (20):
- Germany (20):
  - Charité Berlin, Berlin
  - Elbe Klinikum Buxtehude, Buxtehude
  - Universitätsklinikum Dresden, Dresden
  - HELIOS Klinikum Erfurt, Erfurt
  - Studienzentrum Hautklinik Universitätsklinikum Essen (AöR) Klinik für Dermatologie, Essen
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Medizinische Hochschule Hannover, Hanover
  - Universitätrsklinikum Heidelberg Dermatologie / NCT, Heidelberg
  - SLK Kliniken Heilbronn GmbH, Heilbronn
  - Universitäts-Hautklinik Kiel Klinik f. Dermatologie, Venerologie u. Allergologie, Kiel
  - Universitätsklinikum Leipzig Klinik u. Poliklinik f. Dermatologie, Venerologie u. Allergologie, Leipzig
  - Klinikum der Stadt Ludwigshafen, Ludwigshafen
  - UKSH Campus Lübeck, Lübeck
  - Universitätsklinikum Mainz Hautklinik und Polklinik, Mainz
  - Klinik für Dermatologie, Venerologie und Allergologie UMM - Universitätsmedizin Mannheim, Mannheim
  - Johannes Wesling Klinikum Minden Hautklinik, Minden
  - Universitätsklinikum München (LMU), München
  - Fachklinik Hornheide, Münster
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätshautklinik Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Livingstone E, Zimmer L, Hassel JC, Fluck M, Eigentler TK, Loquai C, Haferkamp S, Gutzmer R, Meier F, Mohr P, Hauschild A, Schilling B, Menzer C, Kiecker F, Dippel E, Roesch A, Ziemer M, Conrad B, Korner S, Windemuth-Kieselbach C, Schwarz L, Garbe C, Becker JC, Schadendorf D; Dermatologic Cooperative Oncology Group. Adjuvant nivolumab plus ipilimumab or nivolumab alone versus placebo in patients with resected stage IV melanoma with no evidence of disease (IMMUNED): final results of a randomised, double-blind, phase 2 trial. Lancet. 2022 Oct 1;400(10358):1117-1129. doi: 10.1016/S0140-6736(22)01654-3. Epub 2022 Sep 10. PMID 36099927
- [Derived] Zimmer L, Livingstone E, Hassel JC, Fluck M, Eigentler T, Loquai C, Haferkamp S, Gutzmer R, Meier F, Mohr P, Hauschild A, Schilling B, Menzer C, Kieker F, Dippel E, Rosch A, Simon JC, Conrad B, Korner S, Windemuth-Kieselbach C, Schwarz L, Garbe C, Becker JC, Schadendorf D; Dermatologic Cooperative Oncology Group. Adjuvant nivolumab plus ipilimumab or nivolumab monotherapy versus placebo in patients with resected stage IV melanoma with no evidence of disease (IMMUNED): a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2020 May 16;395(10236):1558-1568. doi: 10.1016/S0140-6736(20)30417-7. PMID 32416781